CLINICAL TRIAL: NCT04409847
Title: COVID-19 Blood Pressure Endothelium Interaction Study
Brief Title: COVID-19 Blood Pressure Endothelium Interaction Study (OBELIX)
Acronym: OBELIX
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN20CA245
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2021-02

CONDITIONS: COVID; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine samples for vascular phenotpying marker, immuno phenotyping markers and future biomarker studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID+ PCR: Subjects who are SARS-CoV-2 PCR+ve and/or have diagnostic CXR or CT chest features of COVID -19
  Interventions: Diagnostic Test: ABPM; Diagnostic Test: ECG; Diagnostic Test: FMD; Diagnostic Test: PWV; Diagnostic Test: Rarefaction
- COVID- PCR: subjects admitted with COVID-19 like symptoms but are SARS-CoV-2 PCR-ve and have CXR or CT chest that show low probability of COVID-19 will form the control group
  Interventions: Diagnostic Test: ABPM; Diagnostic Test: ECG; Diagnostic Test: FMD; Diagnostic Test: PWV; Diagnostic Test: Rarefaction

INTERVENTIONS:
Diagnostic Test: ABPM — 24 hour ambulatory blood pressure monitoring
Diagnostic Test: ECG — Electrocardiogram
Diagnostic Test: FMD — Flow mediated dilatation
Diagnostic Test: PWV — Pulse wave velocity
Diagnostic Test: Rarefaction — nailbed capillaroscopy

SUMMARY:
The current COVID-19 pandemic (caused by the SARS-CoV-2 virus) represents the biggest medical challenge in decades. Whilst COVID-19 mainly affects the lungs it also affects multiple organ systems, including the cardiovascular system. There are documented associations between severity of disease and risk of death and To provide all the information required by review bodies and research information systems, we ask a number of specific questions. This section invites you to give an overview using language comprehensible to lay reviewers and members of the public. Please read the guidance notes for advice on this section.

5 DRAFT Full Set of Project Data IRAS Version 5.13 advancing age, male sex and associated comorbid disease (hypertension, ischaemic heart disease, diabetes, obesity, COPD and cancer). The most common complications include cardiac dysrhythmia, cardiac injury, myocarditis, heart failure, pulmonary embolism and disseminated intravascular coagulation.

It is thought that the mechanism of action of the virus involves binding to a host transmembrane enzyme (angiotensin- converting enzyme 2 (ACE2)) to enter some lung, heart and immune cells and cause further damage. While ACE2 is essential for viral invasion, it is unclear if the use of the common antihypertensive drugs ACE inhibitors or angiotensin receptor blockers (ARBs) alter prognosis.

This study aims to look closely at the health of the vascular system of patients after being treated in hospital for COVID-19 (confirmed by PCR test) and compare them to patients who had a hospital admission for suspected COVID-19 (negative PCR test) . Information from this study is essential so that clinicians treating patients with high blood pressure understand the impact of the condition and these hypertension medicines in the context of the current COVID-19 pandemic. This will allow doctors to effectively treat and offer advice to patients currently prescribed these medications or who are newly diagnosed with hypertension.

DETAILED DESCRIPTION:
COVID-19 is pandemic and, though it primarily affects the lungs, there is evidence of cardiovascular system involvement. Mechanistically, SARS-CoV-2, following proteolytic cleavage of its S protein by a serine protease, binds to the transmembrane angiotensin-converting enzyme 2 (ACE2) -a homologue of ACE-to enter type 2 pneumocytes, macrophages, perivascular pericytes, and cardiomyocytes. This may lead to myocardial dysfunction and damage, endothelial dysfunction, microvascular dysfunction, plaque instability, and myocardial infarction. While ACE2 is essential for viral invasion, it is unclear if the use of the common antihypertensive drugs ACE inhibitors or angiotensin receptor blockers alter prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Admission between 01/04/2020 and 31/12/2020 Clinically suspected or PCR confirmed COVID-19 Age 30-60 years No history of hypertension or current drug treatment for hypertension

Exclusion Criteria:

* Inability to give informed consent/lack of capacity Non-English speakers BMI >40 eGFR <60 ml/min Pregnancy History of Cancer within 5 years Persistent atrial fibrillation Severe illness, at investigator discretion Prescription of BP lowering drugs Corticosteroid (chronic use) Immunosupressive agents NSAIDs (chronic use)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients admitted through QEUH immediate assessment unit and acute receiving units with suspected or confirmed COVID-19 during 01/04/20 - 31/12/20 and who are alive at discharge. Clinically suspected COVID-19 should have at least two of the following presenting features (fever, new onset cough, fatigue, myalgia, breathlessness, GI symptoms, anosmia/dysgeusia, contact with known COVID-19 positive patient).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
ABPM systolic blood pressure | 24 hours (all day and night)
  Ambulatory Blood Pressure Monitoring systolic blood pressure

SECONDARY OUTCOMES:
24-hr ABPM DBP | 24 hours (all day and night)
  Ambulatory Blood Pressure Monitoring diastolic blood pressure
day ABPM SBP | 8am to 8pm
  Day Ambulatory Blood Pressure Monitoring systolic blood pressure
day ABPM DBP | 8am to 8pm
  Day Ambulatory Blood Pressure Monitoring diastolic blood pressure
night ABPM SBP | 8pm to 8am
  Night Ambulatory Blood Pressure Monitoring systolic blood pressure
night ABPM DBP | 8pm to 8am
  Night Ambulatory Blood Pressure Monitoring diastolic blood pressure
dipping status | 24 hours (all day and night)
  The fall in pressure, called the "dip", is defined as the difference between daytime mean systolic pressure and nighttime mean systolic pressure expressed as a percentage of the day value
morning surge | 24 hours (all day and night)
  he morning surge was defined as the difference between the mean systolic blood pressure during the 2 hours after waking and arising minus the mean systolic blood pressure during the hour that included the lowest blood pressure during sleep.
24 hour ABPM HR | 24hr (all day and night)
  24 hour Ambulatory Blood Pressure Monitoring heart rate
day ABPM HR | 8 am to 8 pm
  Day Ambulatory Blood Pressure Monitoring heart rate
night ABPM HR | 8pm to 8 am
  Night Ambulatory Blood Pressure Monitoring heart rate
Immune phenotyping | at baseline
  Immune phenotyping includes cellular and humoral markers of immune cell activation and senescence within populations of key leukocyte subsets e.g. lymphocytes and monocytes
Microparticle assessments | at baseline
  microparticles are being assessed as biomarkers and biovectors of vascular damage and endothelial dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided